CLINICAL TRIAL: NCT01195701
Title: Clitoral Location in Relation to Sexual Function Using Pelvic MRI: A Case-Control Study
Brief Title: Clitoral Location in Relation to Sexual Function Using Pelvic Imaging
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Collaborators: TriHealth Hatton Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 10063
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Female Sexual Dysfunction; Anorgasmia
Keywords: female sexual dysfunction; anorgasmia; clitoral complex; pelvic MRI; testosterone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood hormone levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Anorgasmia (cases): Women with difficulty or inability to reach sexual climax will be the cases in this study.
- Normal orgasmic function: Women who report that they usually or always achieve sexual climax will be the controls in this study.

SUMMARY:
Women who are unable to achieve orgasm compared to women who have normal orgasmic function may have different clitoral anatomy and different hormone levels. The investigators hypothesis is that women who have difficulty with orgasm may have a clitoris that is closer to the vagina and may have higher testosterone levels. Pelvic MRI will be used to observe whether clitoral measurements differ between women with normal orgasmic function vs. those with anorgasmia.

DETAILED DESCRIPTION:
Women unable with anorgasmia and those with normal orgasmic function will undergo pelvic MRI so that clitoral measurements can be taken and then compared for differences.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female aged 18-55 years
* Sexually active (at least 1 heterosexual partner in the past 4 weeks)
* Cases must have difficulty with orgasm or be anorgasmic
* Controls must have normal sexual function

Exclusion Criteria:

* Not sexually active
* Homosexual orientation
* Postmenopausal
* Stage >2 pelvic organ prolapse (POP-Q measurements beyond hymen)
* Urinary incontinence with coitus limiting sexual activity
* Severe vaginal atrophy
* Pelvic pain/dyspareunia (
* Currently pregnant
* Depression being treated with SSRIs (depression alone or treatment of depression with non-SSRI medications is not an exclusion)
* Currently taking testosterone supplements
* History of sexual abuse
* Large pelvic mass (benign or cancerous) impeding MRI measurements or grossly abnormal pelvic anatomy.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sexually active premenopausal females aged 18-55 years old presenting to private gynecology practice
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Vaccaro, DO, Principal Investigator — Good Samaritan Hospital
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Started | 10 | 25
Completed | 10 | 20
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Population: A sample size calculation determined that with an alpha level of 0.05 a sample size of 13 participants in each arm (N=26) would yield 90% power to detect a mean difference of 5.6 between groups on the FSFI Orgasm subscale. We planned to enroll 40 patients (20 in each arm) to accommodate a predicted dropout rate of approximately 40%.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (8.2) | 31.6 (7.2) | 31.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 19 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clitoral Measurements Using Pelvic MRI
Description: All cases and controls will undergo a pelvic MRI without contrast to assess the clitoral complex.
Time Frame: Between day 1-14 (follicular phase) of menstrual cycle
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
millimeters (mm)
  Glans distance, sagittal, mm | 51.3 (7.6) | 45.1 (5.7)
  Body distance, sagittal, mm | 29.4 (6.8) | 20.6 (3.2)
  Crura distance, medial axial, mm | 24.2 (5.2) | 28.3 (4.6)
  Crura distance, lateral axial, mm | 15.6 (6.1) | 23.8 (3.7)
  Total vaginal length, mm | 84.5 (11.1) | 94.9 (6.5)
  Clitoris to skin distance, mm | 26.6 (11.4) | 27.0 (6.2)
  Midurethra-midvagina distance, mm | 13.3 (2.5) | 12.6 (1)

2. Secondary Outcome: Free Testosterone
Description: Free testosterone and the calculated free androgen index will be compared; additionally, these levels will be correlated with the questionnaire data and clitoral measurements
Time Frame: Between day 1-14 (follicular phase) of menstrual cycle
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
pg/mL | 2.6 [1.9 to 4.6] | 2.5 [2.2 to 3.7]

3. Secondary Outcome: Total Testosterone
Description: Free & total testosterone, and the calculated free androgen index will be compared; additionally, these levels will be correlated with the questionnaire data and clitoral measurements
Time Frame: Between day 1-14 (follicular phase) of menstrual cycle
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
ng/dL | 26.5 [18.2 to 53.2] | 33.0 [28.6 to 43.9]

4. Secondary Outcome: Free Androgen Index
Description: Free androgen index is calculated as the ratio of total testosterone to sex hormone binding globulin (SHBG)
Time Frame: Between day 1-14 (follicular phase) of menstrual cycle
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
ratio | 1.3 [0.9 to 2.4] | 1.2 [1.0 to 1.8]

5. Secondary Outcome: Female Sexual Function Index (FSFI) Total Score
Description: The FSFI is a validated index of sexual function, consisting of a total score and six subscales or domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. The FSFI total is the sum of the six domain scores, each of which is weighted as noted. The FSFI total score can range from 2 to 36, with higher scores indicating better sexual function. A total score of 26.55 has been identified as the ideal cut point for differentiating between normal sexual function and sexual dysfunction.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 20.2 (4.4) | 31.6 (2.7)

6. Secondary Outcome: FSFI Desire
Description: The desire domain of the Female Sexual Function Index (FSFI) consists of two questions and measures the frequency (almost never to almost always) and level (very low to very high) of sexual desire. Item scores range from 1 to 5, with higher scores indicating better sexual function, and the domain score is weighted by a factor of 0.6, such that the domain score can range from 1.2 to 6.0.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 2.6 (1.4) | 4.8 (0.7)

7. Secondary Outcome: FSFI Arousal
Description: The arousal domain of the Female Sexual Function Index (FSFI) consists of four questions and measures the frequency (almost never to almost always) and level (very low to very high) of sexual arousal; and confidence in becoming aroused (very low to very high confidence) and frequency of satisfaction with arousal (almost never to almost always). Item scores range from 0 to 5, with higher scores indicating better sexual function, and the arousal score is weighted by a factor of 0.3, such that the domain score can range from 0 to 6.0.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 3.2 (0.7) | 5.4 (0.6)

8. Secondary Outcome: FSFI Lubrication
Description: The lubrication domain of the Female Sexual Function Index (FSFI) consists of four questions and measures the frequency of lubrication (almost never to almost always), the difficulty in becoming lubricated (extremely difficult to not difficult), frequency of maintaining lubrication (almost never to almost always), and difficulty in maintaining lubrication (extremely difficult to not difficult). Item scores range from 0 to 5, with higher scores indicating better sexual function, and the lubrication score is weighted by a factor of 0.3, such that the domain score can range from 0 to 6.0.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 4.0 (1.3) | 5.5 (0.5)

9. Secondary Outcome: FSFI Orgasm
Description: The orgasm domain of the Female Sexual Function Index (FSFI) consists of three questions and measures the frequency of orgasm (almost never to almost always), difficulty in achieving orgasm (extremely difficult to not difficult), and satisfaction with the ability to reach orgasm (very dissatisfied to very satisfied). Item scores range from 0 to 5, with higher scores indicating better sexual function, and the orgasm score is weighted by a factor of 0.4, such that the domain score can range from 0 to 6.0.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 1.9 (0.7) | 5.6 (0.6)

10. Secondary Outcome: FSFI Satisfaction
Description: The satisfaction domain of the Female Sexual Function Index (FSFI) consists of three questions and measures satisfaction (very dissatisfied to very satisfied) with emotional closeness with partner, sexual relationship with partner, and overall sexual relationship with partner. Item scores range from 0 (or 1) to 5, with higher scores indicating better sexual function, and the satisfaction score is weighted by a factor of 0.4, such that the domain score can range from 0.8 to 6.0.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 3.6 (1.3) | 4.8 (0.8)

11. Secondary Outcome: FSFI Pain
Description: The pain domain of the Female Sexual Function Index (FSFI) consists of three questions and measures the frequency of discomfort or pain during and following vaginal penetration (almost never to almost always), and the level of discomfort or pain (very low to very high). Item scores range from 0 to 5, with higher scores indicating better sexual function, and the pain score is weighted by a factor of 0.4, such that the domain score can range from 0 to 6.0.
Time Frame: baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Number analyzed (Participants) | 10 | 20
units on a scale | 4.9 (1.1) | 5.5 (0.6)

ADVERSE EVENTS:
Arm/Group | Anorgasmia (Cases) | Normal Orgasmic Function
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No